CLINICAL TRIAL: NCT06173011
Title: A Randomized, Double-blind, Single-dose, Parallel Three-group Study to Compare the Pharmacokinetics and Safety of QL2107 and Keytruda® (Marketed in China and the United States) in Healthy Male Adults
Brief Title: A Study Comparing Pharmacokinetic and Safety of QL2107 and Keytruda® (Marketed in China and the United States) in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2107-101
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QL2107 (Experimental): QL2107, intravenous infusion 35 min (±5min, minimum infusion 30min), D1 (Day 1, single dose)
  Interventions: Drug: QL2107
- Keytruda®(china) (Active Comparator): Keytruda® (china), intravenously infusion 35 min (±5min, at least 30min), D1 (Day 1, single dose);
  Interventions: Drug: Keytruda®(china)
- Keytruda®(US) (Active Comparator): Keytruda® (US), intravenously infusion 35 min (±5min, at least 30min), D1 (Day 1, single dose);
  Interventions: Drug: Keytruda®(US)

INTERVENTIONS:
Drug: QL2107 — intravenous infusion 35 min (±5min, minimum infusion 30min), D1 (Day 1, single dose)
  Arms: QL2107
Drug: Keytruda®(china) — intravenous infusion 35 min (±5min, minimum infusion 30min), D1 (Day 1, single dose)
  Arms: Keytruda®(china)
Drug: Keytruda®(US) — intravenous infusion 35 min (±5min, minimum infusion 30min), D1 (Day 1, single dose)
  Arms: Keytruda®(US)

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic and safety similarity of QL2107 with Keytruda® marketed in China and the United States in healthy male volunteers.

Participants will receive a single injection of QL2107/ Keytruda® （China）/Keytruda® （US）.Researchers will compare pharmacokinetic, safety, and immunogenic similarities between the three groups.

DETAILED DESCRIPTION:
This is a phase I,single center, randomized, double-blind and parallel group clinical trial .

The primary objective is to assess the pharmacokinetic similarity of single injections of QL2107 or Keytruda® （China/US） in healthy volunteers.

The secondary objective are to assess the clinical safety and immunogenicity similarity of single injections of QL2107 or Keytruda® （China/US） in healthy volunteers.

Subjects would receive a single 100mg（4ml） of QL2107or Keytruda® （China/US）injection.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
2. Age 18 ~ 50 (inclusive) years , male;
3. 50.0 kg≤ body weight ≤90.0 kg and 18.0 kg/m2≤ Body mass index (BMI) ≤28.0 kg/m2;
4. Agree to use effective contraception throughout the study period (including but not limited to: physical contraception, surgery, abstinence, etc.) until at least 6 months after the study dosing;
5. No history of disease or abnormal past medical history is not clinically significant, and the study doctor's judgment has no impact on the trial.

Exclusion criteria

Exclusion Criteria:

1. Clinical laboratory examination, infectious disease screening, chest orthogram examination, abdominal color ultrasound examination, 12-lead electrocardiogram, heart color ultrasound, physical examination, vital signs (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg) the abnormalities in each examination have clinical significance or are determined to have an impact on the trial (subject to the judgment of the clinical study physician);

(2) Have been or are currently suffering from any clinically serious disease of the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatric and metabolic abnormalities, or any other disease that can interfere with the test results;

3. Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to: rheumatoid arthritis, ankylosing spondylitis, autoimmune hemolytic anemia, interstitial pneumonia, uveitis, inflammatory bowel disease, autoimmune hepatitis, autoimmune pituitaritis, glomerulonephritis, hyperthyroidism or hypothyroidism, etc.)

4. Known history of tuberculosis or suspected clinical manifestations of tuberculosis (including but not limited to tuberculosis, lymphatic tuberculosis, tuberculous pleurisy, etc.);

5. Patients with a history of acute infection within 2 weeks before screening;

6. There have been herpes zoster virus infections within 3 months before screening;

7. Viral hepatitis (including hepatitis B and C), AIDS antibody, treponema pallidum antibody screening positive;

8. Allergies (multiple drug and food allergies), who were determined by the researcher to be unable to participate in this study;

9. Patients who had surgery within 4 weeks prior to screening or planned to have surgery during the study period;

10. Those who have used any biological product or received live viral vaccine (tetanus toxoid vaccine within 1 year before infusion), used any monoclonal antibody within 6 months or 5 biological half-lives of drug metabolism, or used PD-1/PD-L1 drugs in the past;

11. Those who have used any drug or health product (including Chinese herbal medicine) within 14 days prior to the infusion of the experimental drug;

12. Participants who participated in any clinical trial and used any clinical trial drug within 3 months prior to screening;

13. Study patients who donated blood or lost a large amount of blood (> 400 mL) or received blood transfusions or used blood products within 3 months prior to administration;

14. Smokers or smokers who smoked more than 5 cigarettes per day in the 3 months prior to screening or who could not stop using any tobacco products during the trial;

15. Positive drug screening or/and alcohol breath test screening prior to study administration;

16. A history of drug and/or alcohol abuse (14 units of alcohol consumed per week "1 unit = 285 mL for beer, 25 mL for spirits, or 100 mL for wine");

17. Subjects who have other factors deemed unsuitable for the study by the investigator;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda® (china/US)after a single intravenous infusion in healthy volunteers

SECONDARY OUTCOMES:
safety and immunogenicity | 113day
  Safety, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0.after a single intravenous infusion in healthy volunteers;Immunogenicity will be assessed by the incidence of ADA and Nab.
Cmax | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
Tmax | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
AUC0-t | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
t1/2 | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
CL | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
Vd | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®
AUC_%Extrap | 113day
  To evaluate pharmacokinetic similarity between QL2107 and Keytruda®

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jilin University, Changchun, Jilin, China